CLINICAL TRIAL: NCT07196618
Title: Effect of Dimethyl Sulfoxide Pretreatment on Tensile Bond Strength and Nanoleakage of Resin Composite Bonded to Aged Dentin
Brief Title: Bond Strength Evaluation
Acronym: DMSO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Aisha Nasr Ali Zahran, Doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P-OP-23-03
Record Dates: First submitted 2025-08-09; First posted 2025-09-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Bonding
MeSH Terms: interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DMSO (Active Comparator)
  Interventions: Drug: dimethyl sulfoxide
- CHX (Active Comparator)
  Interventions: Drug: Cholorhexidine

INTERVENTIONS:
Drug: dimethyl sulfoxide — dentin pretreated using dimethyl sulfoxide and follow up of patients at 2 weeks, 3 months and 6 months
  Arms: DMSO
Drug: Cholorhexidine — dentin pretreated using chlorhexidine and follow up of patients at 2 weeks, 3months and 6 months
  Arms: CHX

SUMMARY:
This study was evaluated the effect of dimethyl sulfoxide pretreatment on tensile bond strength and nanoleakage of resin composite bonded to aged dentin.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study will be required to present at least one of non caries cervical lesion with sclerotic dentin without pulpal involvement.
* Age of patient: 50 - 75 years
* Patients with non caries cervical lesion will be standardized by clinical performance (FDI world dental federation).

Exclusion Criteria:

* Teeth with deep dentinal lesions with pulpal involvement, abscess, pain or swelling
* Developmental disorders and adjacent soft tissue lesions
* Patients with systemic illness will be excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
clinical assessment evaluation using the FDI world dental federation criteria | post operative 2 weeks

SECONDARY OUTCOMES:
clinical assessment evaluation using the FDI world dental federation criteria | post operative 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Zahran, Study Director — Al-Azhar University
Locations (1):
- Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No